CLINICAL TRIAL: NCT06095960
Title: Comparative Evaluation of Telehealth Multi-Component Optional Model (MOM) of Postpartum Care Among Rural, Low-income, and Diverse Women
Brief Title: Telehealth Multi-Component Optional Model (MOM) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 276311
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Maternal Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth MOM (Experimental): Telehealth MOM. Each patient will receive ESoC which includes: education on the symptoms to watch for and when to call their healthcare provider, an in-person comprehensive postpartum visit around 6 weeks postpartum, and any additional care deemed necessary by their health care providers. Patients in the Telehealth MOM arm will be also provided with a remote monitoring blood pressure cuff and thermometer and will be instructed to take their blood pressure and temperature twice a day for 14 days after discharge from the hospital. A Registered Nurse will monitor blood pressure and temperature readings over the 14-day period and will contact the patient if the readings are out of range to discuss symptoms and the recommend a course of action. A Registered Nurse will conduct an early postpartum telehealth visit between 10-14 days postpartum.
  Interventions: Behavioral: Telehealth MOM
- Enhanced Standard of Care (Active Comparator): Enhanced standard of care (ESoC). Each patient will be provided education on the symptoms to watch for and when to call their healthcare provider. Patients will be scheduled for a comprehensive postpartum visit around 6 weeks postpartum and any additional care deemed necessary by their health care providers.
  Interventions: Other: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: Telehealth MOM — Patients will receive enhanced standard of care plus remote blood pressure monitoring, remote thermometer, and a 10- to 14-day post-partum telehealth visit.
  Arms: Telehealth MOM
Other: Enhanced Standard of Care — Patients will receive enhanced standard of care which includes: education on symptoms and when to call their healthcare provider, comprehensive 6-week post-partum visit, and any healthcare deemed necessary by providers.
  Arms: Enhanced Standard of Care

SUMMARY:
The aim of this study is to conduct a comparative effectiveness evaluation using a randomized control trail design among diverse women to compare two postpartum care models: 1) Telehealth Multicomponent Optimal Model (Telehealth MOM) and 2) enhanced standard of care (ESoC). This study will address critical gaps in knowledge about how best to deliver comprehensive postpartum care that ensures timely identification and treatment of complications and meets the needs and preferences of diverse patients, including disproportionately-impacted racial groups and rural residents.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 16-35 weeks gestation
* Age 18-44 years
* Ability to speak English, Spanish, or Marshallese
* Participants may have either a vaginal birth or cesarean section birth

Exclusion Criteria:

* Type 1 diabetes on an insulin pump followed closely by endocrinology
* Uncontrolled Type 2 diabetes
* End stage renal disease followed closely by nephrology
* ICU admission at any point during pregnancy or delivery hospitalization
* Other maternal conditions requiring additional surgeries (i.e. cesarean hysterectomy or intrapartum or postpartum oophorectomy/appendectomy)
* Incarceration
* Mental disability limiting decision-making capacity
* Uncontrolled chronic hypertension
* HELLP syndrome during pregnancy
* Sickle cell disease
* Maternal heart condition or heart disease
* Opioid use disorder
* Lupus
* Thrombophilia or blood clots
* Need for blood transfusion during delivery hospitalization
* Other maternal conditions or complications, known during pregnancy or delivery hospitalization, requiring prolonged hospitalization postpartum

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Completion of post-partum 6-week comprehensive visit | Baseline to 6 weeks post-partum
  Binary measure (yes/no) of visit completion

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Callaghan-Koru, PhD, Principal Investigator — University of Arkansas; Pearl McElfish, PhD, Principal Investigator — University of Arkansas
Locations (6):
- United States (6):
  - UAMS El Dorado FMC, El Dorado, Arkansas
  - UAMS Fayetteville FMC, Fayetteville, Arkansas
  - UAMS Fort Smith FMC, Fort Smith, Arkansas
  - UAMS Jonesboro FMC, Jonesboro, Arkansas
  - UAMS Health Women's Center, Little Rock, Arkansas
  - UAMS Springdale FMC, Springdale, Arkansas

IPD SHARING:
Plan to Share IPD: No